CLINICAL TRIAL: NCT04683913
Title: Foot Progression Angle Modification: an Exploratory Six-week Telerehabilitation Intervention in People With Knee Osteoarthritis
Brief Title: Telerehabilitation Gait Modification
Acronym: TELEMOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Michael Hunt, Professor, Assoc Dean, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H20-03086
Record Dates: First submitted 2020-12-15; First posted 2020-12-24 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-10

CONDITIONS: Osteoarthritis, Knee
Keywords: Gait Modification; Wearable Sensors; Real-world Monitoring; Telerehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Two-arm delayed control design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention: Telerehabilitation (Experimental): Immediate entry into the gait modification intervention delivered using teleconferencing methods
  Interventions: Behavioral: Foot rotation modification
- Delayed Intervention: Telerehabilitation (Experimental): Delayed (6 weeks) entry into the gait modification intervention delivered using teleconferencing methods
  Interventions: Behavioral: Foot rotation modification; Other: Waiting Period - Delayed Group

INTERVENTIONS:
Behavioral: Foot rotation modification — The instruction of gait modification provided via teleconferencing sessions (5 over 6 weeks) focusing on increasing toe-in or toe-out angles by "as much as is comfortable".
  Other Names: gait modification
Other: Waiting Period - Delayed Group — Participants allocated to the Delayed Group will wait 6 weeks after their initial baseline, then complete a second baseline to provide a control condition. After the second baseline they will enter the intervention.
  Other Names: control
  Arms: Delayed Intervention: Telerehabilitation

SUMMARY:
Excessive knee joint loads during walking can contribute to knee osteoarthritis progression. Changing the rotation of the foot (in-toeing or out-toeing) while walking can lower knee joint loads and improve pain and function. Telerehabilitation (using video or telephone communication to delivery rehabilitation) has shown promise in delivering exercise therapy for knee osteoarthritis, but it is unknown if walking modifications can be delivered using this method. This study consists of a six-week walking modification program in people with knee osteoarthritis. Performance of the modification will be measured using motion capture and wearable sensors during practice and daily life.

DETAILED DESCRIPTION:
Loads on the knee joint during walking are related to worsening of knee osteoarthritis. Changing walking motions to lower these knee joint loads is an emerging management strategy for knee osteoarthritis. Multiple studies have targeted a change in the position of the foot relative to the direction of walking (toe-in or toe-out walking) and have shown this walking modification to lower knee joint loads and improve symptoms (e.g. pain) related to knee osteoarthritis within the context of a walking program. Building off the many studies that have found telerehabilitation to be an effective method of providing exercise and pain-coping physical therapy, the investigators will use this method to provide walking modification treatment. Telerehabilitation (using video or teleconferencing to conduct the physical therapy appointment) provides a convenient and cost-effective method to work with patients and coordinate their treatment plan. To monitor progress with learning the walking modification, the investigators will use a custom sensor shoe that the participants will wear during daily walking activities over the six-week intervention. Overall, this study will investigate the feasibility and effectiveness of a walking modification program delivered using video- or teleconference.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older
* Exhibit signs of tibiofemoral osteoarthritis based on a score of ≥2 on the Kellgren and Lawrence grading scale predominantly in the medial compartment.
* Self-reported knee pain ≥ 3 / 10 on a numerical rating scale of pain (NRS; 0 = "no pain" and 10 = "worst pain imaginable") during most days of the previous month
* Comfortable walking intermittently for 30 minutes
* Fit into the available sizes of sensor shoes (between US women's 5 to men's 13)
* Exhibits ≥2% reduction in knee adduction moment impulse at 10 degrees of change in toe-in or toe-out during the screening appointment.

Exclusion Criteria:

* Any knee surgery or intraarticular injections within the past 6 months
* A history of joint replacement surgery or high tibial osteotomy
* Current or recent (within 6 weeks) corticosteroid injections
* Use of a gait aid
* Currently on a wait list for joint replacement surgery or high tibial osteotomy
* Any inflammatory arthritic condition
* Any other conditions that may affect normal gait or participation in an aerobic exercise program
* Cannot attend all required appointments

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Motion Analysis and Biofeedback Laboratory, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two recruitment drives were completed using online social media outlets between January 2021 and May 2021. The drives garnered 134 respondents (72 and 62, respectively) who were preliminarily screened for study inclusion/exclusion. Sixty individuals underwent radiographic screening and 28 underwent biomechanical screening for response to gait modification. A total of 20 participants completed baseline assessments and were randomized.
Pre-assignment Details: Participants completed a biomechanical screen involving normal and modified walking in a motion capture space. The data were used to calculate the knee adduction moment impulse (main biomechanical outcome) and foot progression angle (modification target). Those who did not reduce their knee adduction moment impulse >5% were not included in the study.
Period: Overall Study
Arm/Group | Immediate Intervention: Telerehabilitation | Delayed Intervention: Telerehabilitation
Started | 10 | 10
Baseline | 10 | 10
Follow up | 10 | 10
Secondary Baseline | 0 | 10
Retention | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Intervention: Telerehabilitation | Delayed Intervention: Telerehabilitation | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (7.2) | 67.9 (3.2) | 67.4 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 1 | 2 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 10 | 10
Height [Mean (Standard Deviation); unit: cm] | 167.3 (9.6) | 169.3 (9.1) | 168.3 (9.1)
Body Mass [Median (Standard Deviation); unit: kg] | 75.7 (18.1) | 75.2 (11.7) | 75.4 (14.9)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.8 (4.7) | 26.2 (3.8) | 26.5 (4.2)
Knee Symptom Laterality [Count of Participants; unit: Participants]
  Bilateral | 9 | 5 | 14
  Unilateral | 1 | 5 | 6
Symptom Duration [Mean (Standard Deviation); unit: months] | 114.3 (72.0) | 80.2 (78.3) | 97.2 (75.2)
Kellgren and Lawrence Grade [Count of Participants; unit: Participants] — The Kellgren and Lawrence grading scale was used to quantify the severity of structural signs of osteoarthritis in the knee. The scale ranges from 0 to 4 with 0 representing no signs of osteoarthritis and 4 representing severe osteoarthritis. Grading was performed by two experienced team members (over 30 years combined experience) and the final score was based on consensus.
  Participants
    Kellgren and Lawrence 2 | 4 | 3 | 7
    Kellgren and Lawrence 3 | 3 | 4 | 7
    Kellgren and Lawrence 4 | 3 | 3 | 6
Foot Progression Angle Direction Prescription [Count of Participants; unit: Participants]
  Toe-in | 6 | 5 | 11
  Toe-out | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Lab-measured Performance of Gait Modification
Description: Change in foot rotation angle between baseline and week 6 (follow-up) appointments measured using marker-based motion capture. Foot rotation is defined as the angle between the long axis of the foot and the walking direction. Measures of central tendency and variability will be extracted.
Time Frame: Baseline, Week 6
Measure: Mean (95% Confidence Interval); unit: degrees
Arm/Group | Immediate Intervention: Telerehabilitation | Delayed Intervention: Telerehabilitation
Number analyzed (Participants) | 10 | 10
degrees
  Baseline | 6.32 [4.25 to 8.40] | 5.71 [3.03 to 8.39]
  Week 6 | 11.22 [7.0 to 15.43] | 5.64 [2.90 to 8.38]
Statistical Analysis 1: Comparison: Immediate Intervention: Telerehabilitation vs Delayed Intervention: Telerehabilitation; Test type: Other; p < 0.001, ANCOVA; alpha=0.05

2. Primary Outcome: Real-world Performance of Gait Modification
Description: Change in absolute median foot rotation from baseline to each real-world walking bout (represented as a single data file on the sensor module), follow-up, and retention measured via the sensor shoe. Foot rotation is defined as the angle between the long axis of the foot and the walking direction. Measures of central tendency and variability will be extracted, in addition to the proportion of steps with a greater than or equal to 7 degree change.
Time Frame: Baseline, Week 1&2, Week 3&4, Week 5&6, Follow up (Week 6/12), Retention (Week 10/16)
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Delayed Intervention: Telerehabilitation: Delayed (6 weeks) entry into the gait modification intervention delivered using teleconferencing methods Foot rotation modification: The instruction of gait modification provided via teleconferencing sessions (5 over 6 weeks) focusing on increasing toe-in or toe-out angles by "as much as is comfortable".
  Waiting Period - Delayed Group: Participants allocated to the Delayed Group will wait 6 weeks after their initial baseline, then complete a second baseline to provide a control condition. After the second baseline they will enter the intervention.
- Immediate Intervention: Telerehabilitation: Immediate entry into the gait modification intervention delivered using teleconferencing methods Foot rotation modification: The instruction of gait modification provided via teleconferencing sessions (5 over 6 weeks) focusing on increasing toe-in or toe-out angles by "as much as is comfortable".
Arm/Group | Delayed Intervention: Telerehabilitation | Immediate Intervention: Telerehabilitation
Number analyzed (Participants) | 10 | 10
degrees
  Week 1&2 | 8.0 (7.1) | 5.3 (3.9)
  Week 3&4 | 10.8 (6.7) | 9.26 (3.4)
  Week 5&6 | 12.0 (6.6) | 7.7 (4.4)
  Follow up | 11.9 (6.6) | 10.9 (4.6)
  Retention | 5.9 (3.2) | 9.73 (4.5)
Statistical Analysis 1: Comparison: Delayed Intervention: Telerehabilitation; The change in foot progression angle magnitude at each sequential time point were compared using paired t-tests (with a Bonferroni-Dunn correction). Results indicate whether the change from baseline were significantly different at each time point. Abbreviations: F=Follow up, R=Retention; Test type: Other; p = 0.027, t-test, 2 sided — Week 1&2 vs Week 3&4; alpha corrected with Bonferroni-Dunn procedure (k=10)
Statistical Analysis 2: Comparison: Delayed Intervention: Telerehabilitation; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 1.0, t-test, 2 sided — Week 3&4 vs Week 5&6
Statistical Analysis 3: Comparison: Delayed Intervention: Telerehabilitation; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.078, t-test, 2 sided — Week 5&6 vs Follow up; alpha corrected with Bonferroni-Dunn procedure (k=10)
Statistical Analysis 4: Comparison: Delayed Intervention: Telerehabilitation; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.015, t-test, 2 sided — Follow up vs Retention; alpha corrected with Bonferroni-Dunn procedure (k=10)
Statistical Analysis 5: Comparison: Delayed Intervention: Telerehabilitation; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.567, t-test, 2 sided — Week 1&2 vs Week 5&6; alpha corrected with Bonferroni-Dunn procedure (k=10)
Statistical Analysis 6: Comparison: Delayed Intervention: Telerehabilitation; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.001, t-test, 2 sided — Week 1&2 vs Follow up; alpha corrected with Bonferroni-Dunn procedure (k=10)
Statistical Analysis 7: Comparison: Delayed Intervention: Telerehabilitation; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 1.0, t-test, 2 sided — Week 1&2 vs Retention; alpha corrected with Bonferroni-Dunn procedure (k=10)
Statistical Analysis 8: Comparison: Delayed Intervention: Telerehabilitation; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.205, t-test, 2 sided — Week 3&4 vs Follow up; alpha corrected with Bonferroni-Dunn procedure (k=10)
Statistical Analysis 9: Comparison: Delayed Intervention: Telerehabilitation; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.162, t-test, 2 sided — Week 3&4 vs Retention; alpha corrected with Bonferroni-Dunn procedure (k=10)
Statistical Analysis 10: Comparison: Delayed Intervention: Telerehabilitation; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.421, t-test, 2 sided — Week 5&6 vs Retention; alpha corrected with Bonferroni-Dunn procedure (k=10)

3. Primary Outcome: Intervention Adherence
Description: Adherence will be measured by the ratio of telerehabilitation sessions the participant attends relative to the total sessions (5 total).
Time Frame: Week 6
Measure: Mean (Full Range); unit: percent of sessions attended
Arm/Group | Delayed Intervention: Telerehabilitation | Immediate Intervention: Telerehabilitation
Number analyzed (Participants) | 10 | 10
percent of sessions attended | 100 [100 to 100] | 100 [100 to 100]

4. Primary Outcome: Compliance With Gait Modification
Description: Compliance will be estimated by self-reported confidence in performing the gait modification (where 0 = "no confidence" and 10 = "complete confidence") at follow up. Acceptable confidence ratings by week 6 are greater than or equal to 7/10.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Delayed Intervention: Telerehabilitation | Immediate Intervention: Telerehabilitation
Number analyzed (Participants) | 10 | 10
score on a scale | 8.7 (1.3) | 8.4 (1.3)

5. Primary Outcome: Difficulty in Performing the Modification
Description: Difficulty of performing the modification at week 6. Difficulty measured on an NRS scale (0 = no difficulty and 10 = most difficulty possible). Acceptable difficulty by week 6 is less than or equal to 4/10.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Delayed Intervention: Telerehabilitation | Immediate Intervention: Telerehabilitation
Number analyzed (Participants) | 10 | 10
score on a scale | 1.9 (1.7) | 2.0 (1.6)

6. Primary Outcome: Satisfaction With the Treatment Program
Description: Satisfaction with the gait modification program on a 7-point Likert scale where -3 = "extremely unsatisfied" and +3 = "extremely satisfied". Scores of +2 or +3 will be considered "satisfied" and acceptable.
Time Frame: Week 6
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Delayed Intervention: Telerehabilitation | Immediate Intervention: Telerehabilitation
Number analyzed (Participants) | 10 | 10
score on a scale | 2.5 [1 to 3] | 2 [2 to 3]

7. Secondary Outcome: Knee-osteoarthritis Related Symptoms
Description: Change in pain (9 items), stiffness (7 items), physical function (17 items), and quality of life (4 items) will be measured by the Knee Injury and Osteoarthritis Outcome Score at baseline, follow up and retention. Each item is rated on a 5 points Likert scale where 0 = "No problems" and 4 = "Extreme Problems". Higher scores indicate better function. The scores are normalized to 0-100%.
Time Frame: Baseline, Week 6
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Immediate Intervention: Telerehabilitation | Delayed Intervention: Telerehabilitation
Number analyzed (Participants) | 10 | 10
scores on a scale
  Baseline Pain | 60.6 [50.2 to 70.9] | 59.2 [51.1 to 67.2]
  Week 6 Pain | 65.0 [57.1 to 72.9] | 61.9 [54.9 to 69.0]
  Baseline Stiffness | 55.0 [43.9 to 66.1] | 60.7 [49.1 to 72.3]
  Week 6 Stiffness | 65.0 [57.1 to 72.9] | 61.4 [52.0 to 70.8]
  Baseline Physical Function | 65.9 [53.1 to 78.6] | 72.9 [63.8 to 82.1]
  Week 6 Physical Function | 74.3 [66.7 to 81.8] | 77.6 [68.5 to 86.8]
  Baseline Quality of Life | 41.0 [26.6 to 55.4] | 42.0 [28.8 to 55.2]
  Week 6 Quality of Life | 47.0 [37.3 to 56.7] | 48.5 [33.1 to 63.9]
Statistical Analysis 1: Comparison: Immediate Intervention: Telerehabilitation vs Delayed Intervention: Telerehabilitation; Knee Injury and Osteoarthritis Outcome Scale - pain subscale scores were compared between the delayed and immediate groups at week 6 using ANCOVA; Test type: Superiority; p = 0.750, ANCOVA; Controlling for baseline scores, structural severity and sex. alpha=0.05
Statistical Analysis 2: Comparison: Immediate Intervention: Telerehabilitation vs Delayed Intervention: Telerehabilitation; Knee Injury and Osteoarthritis Outcome Scale - stiffness subscale scores were compared between the delayed and immediate groups at week 6 using ANCOVA; Test type: Superiority; p = 0.201, ANCOVA; Controlling for baseline scores, structural severity and sex. alpha=0.05
Statistical Analysis 3: Comparison: Immediate Intervention: Telerehabilitation vs Delayed Intervention: Telerehabilitation; Knee Injury and Osteoarthritis Outcome Scale - physical function subscale scores were compared between the delayed and immediate groups at week 6 using ANCOVA; Test type: Superiority; p = 0.997, ANCOVA; Controlling for baseline scores, structural severity and sex. alpha=0.05
Statistical Analysis 4: Comparison: Immediate Intervention: Telerehabilitation vs Delayed Intervention: Telerehabilitation; Knee Injury and Osteoarthritis Outcome Scale - quality of life subscale scores were compared between the delayed and immediate groups at week 6 using ANCOVA; Test type: Superiority; p = 0.423, ANCOVA; Controlling for baseline scores, structural severity and sex. alpha=0.05

8. Secondary Outcome: Knee Joint Moments
Description: Peaks and impulse of the knee adduction moment and knee flexion moment measured via in-laboratory gait analysis (force platforms and marker-based motion capture) at baseline, and follow up.
Time Frame: Baseline, Week 6
Measure: Mean (95% Confidence Interval); unit: Nm/kg
Arm/Group | Immediate Intervention: Telerehabilitation | Delayed Intervention: Telerehabilitation
Number analyzed (Participants) | 10 | 10
Nm/kg
  Baseline KAM1 | 0.56 [0.42 to 0.7] | 0.50 [0.39 to 0.6]
  Week 6 KAM1 | 0.49 [0.35 to 0.62] | 0.45 [0.36 to 0.53]
  Baseline KAM2 | 0.30 [0.22 to 0.37] | 0.33 [0.24 to 0.41]
  Week 6 KAM2 | 0.28 [0.18 to 0.38] | 0.32 [0.24 to 0.40]
  Baseline KFM peak | 0.70 [0.58 to 0.81] | 0.66 [0.51 to 0.82]
  Week 6 KFM peak | 0.72 [0.63 to 0.80] | 0.68 [0.53 to 0.83]
Statistical Analysis 1: Comparison: Immediate Intervention: Telerehabilitation vs Delayed Intervention: Telerehabilitation; Knee adduction moment 1 (early stance) was analyzed as raw Nm with body mass entered as as covariate; Test type: Superiority; p = 0.342, ANCOVA; Controlling for body mass, structural severity and sex. alpha=0.05
Statistical Analysis 2: Comparison: Immediate Intervention: Telerehabilitation vs Delayed Intervention: Telerehabilitation; Knee Adduction Moment 2 (late stance was analyzed as raw Nm with body mass entered as as covariate; Test type: Superiority; p = 0.844, ANCOVA; Controlling for body mass, structural severity and sex. alpha=0.05
Statistical Analysis 3: Comparison: Immediate Intervention: Telerehabilitation vs Delayed Intervention: Telerehabilitation; Knee Flexion Moments were analyzed as raw Nm with body mass entered as as covariate; Test type: Superiority; p = 0.774, ANCOVA; Controlling for body mass, structural severity and sex. alpha=0.05

9. Secondary Outcome: Knee Joint Moment Impulse
Description: Impulse of the knee adduction and flexion moments.
Time Frame: Baseline, Week 6
Measure: Mean (95% Confidence Interval); unit: Nm/kg*s
Arm/Group | Immediate Intervention: Telerehabilitation | Delayed Intervention: Telerehabilitation
Number analyzed (Participants) | 10 | 10
Nm/kg*s
  KAM Impulse Baseline | 0.16 [0.12 to 0.20] | 0.18 [0.14 to 0.22]
  KAM Impulse Week 6 | 0.15 [0.11 to 0.18] | 0.17 [0.11 to 0.18]
  KFM Impulse Baseline | 0.1 [0.08 to 0.12] | 0.13 [0.07 to 0.19]
  KFM Impulse Week 6 | 0.11 [0.09 to 0.12] | 0.13 [0.07 to 0.19]
Statistical Analysis 1: Comparison: Immediate Intervention: Telerehabilitation vs Delayed Intervention: Telerehabilitation; Knee adduction moment impulses were analyzed as raw Nm*s with body mass entered as as covariate; Test type: Superiority; p = 0.186, ANCOVA; Controlling for body mass, structural severity and sex. alpha=0.05
Statistical Analysis 2: Comparison: Immediate Intervention: Telerehabilitation vs Delayed Intervention: Telerehabilitation; Knee flexion moment impulses were analyzed as raw Nm*s with body mass entered as as covariate; Test type: Superiority; p = 0.601, ANCOVA; Controlling for body mass, structural severity and sex. alpha=0.05

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the six week intervention period. For the immediate group this was Week 0 to Week 6 and for the delayed group this was Week 6 to Week 12. Adverse events were reported at each telerehabilitation appointment with the study interventionist.
Description: Adverse event data collected by participant self-report. These measures are presented for the whole study sample as the data for the two intervention periods (immediate and delayed groups) were combined for the pre-post analysis in this study.
Arm/Group | Delayed Intervention: Telerehabilitation | Immediate Intervention: Telerehabilitation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 7/10 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed Intervention: Telerehabilitation (N=10) | Immediate Intervention: Telerehabilitation (N=10)
Hip/thigh discomfort (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Knee discomfort (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
Ankle/foot discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT04683913/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT04683913/SAP_001.pdf